CLINICAL TRIAL: NCT02381444
Title: Health Related Quality of Life in LCIG Patients and LCIG Patients and LCIG Eligible Patients Continuing Oral Therapy. A Multicenter Post Marketing Observational Study for LCIG in Germany and Switzerland - BALANCE
Brief Title: Health Related Quality of Life in LCIG Patients and LCIG Eligible Patients Continuing Oral Therapy
Acronym: BALANCE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-322
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Parkinson's Disease (PD)
Keywords: Advanced Parkinson's Disease; Levodopa Carbidopa Intestinal Gel; Observational Study; Quality of life; Jejunal Percutaneous Endoscopic Gastrostomy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard of Care: Participants with advanced Parkinson's Disease
- Levodopa Carbidopa Intestinal Gel: Participants with advanced Parkinson's Disease

SUMMARY:
The aim of this study is to assess the effect of LCIG (levodopa-carbidopa intestinal gel) on HRQL (Health-Related Quality of Life) of participants and compare the Health-Related Quality of Life between participants continuing to levodopa-carbidopa intestinal gel treatments versus participants continuing on oral therapy for Parkinson's Disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disorder in the world. It can be treated sufficiently until motor complications with fluctuations of mobility and dyskinesia develop. The quality of life is relentlessly deteriorating with longer disease duration once the complications of conservative oral therapy develop. Continuous dopaminergic stimulation using Levodopa/Carbidopa Intestinal Gel (LCIG) improves the motor complications of Parkinson's disease and preliminary data suggest that also the quality of life is improved. Primary Objective is to assess the effect of LCIG on Health Related Quality of Life (HRQL) of patients according to selection criteria from German guidelines and compare improvement in HRQL between patients continuing to LCIG treatment and patients staying on oral treatment, despite being eligible according to these guidelines. In addition, current selection criteria recommended by the national guideline will be documented at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for LCIG according to current version of the Summary of Product Characteristics of LCIG of the respective country (Germany, Switzerland).
* Decision to treat with LCIG or other medication made by the study physician prior to any decision to approach the patient to participate in this study.
* Unchanged available combinations of PD medicinal treatment for at least one week prior to study inclusion.
* Patient has given written informed consent.

Exclusion Criteria:

* Contraindication to LCIG according to current version of the German SmPC or Swiss SmPC.
* Contraindication to placement of intrajejunal PEG-J tube.
* Current treatment with Deep Brain Stimulation (DBS), Apomorphine pump or LCIG
* Severe dementia based on a Mini-Mental State Examination (MMSE) of < 10
* Acute psychotic disorder (benign hallucinations or earlier psychotic episodes are not an exclusion criterion)
* Depression with suicidal thoughts (earlier episodes of major depression are not an exclusion criterion)
* History or presence of any condition that might interfere with absorption, distribution, metabolism, or excretion of LCIG
* Drug or alcohol addiction (drug addiction: continuous or sporadic use of drugs without medical indication or with paradoxical medical indication or in inappropriate amounts. Addictive consumption of e.g. alcohol, cannabis, amphetamine, sniffing agents, cocaine, heroin, crack). Alcohol addiction male: > 40 g/day; female: > 30 g/day)
* Illiteracy or insufficient language skills to complete the questionnaires

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Parkinson Disease
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2015-04-17 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Change in the Parkinson's Disease Questionnaire (PDQ-39) summary index | From baseline to 12 months
  The primary endpoint is the change in the Parkinson's Disease Questionnaire (PDQ-39) summary index from 12 months to the baseline assessment. The two treatment groups levodopa-carbidopa intestinal gel vs. Standard of Care will be compared.

SECONDARY OUTCOMES:
Change in Health Related Quality of Life (HRQL) | At Baseline, 6, and 12 months of treatment
  Unified Parkinson's disease Rating Scale (UPDRS) part III in the medication "on" state
Change in participant's motor symptoms | From Baseline to 6 and 12 months of treatment.
  Activities of daily living "on" and "off" medication - Unified Parkinson's disease Rating Scale (UPDRS) part II
Change in participant's Healthcare Resource Utilization | From Baseline to 6 and 12 months of treatment
  Frequency and severity of ON-dyskinesia (Unified Parkinson's Disease Rating Scale part IV, Complications of Therapy: Items 32, 33, 34 and 39)
Change in participant's non-motor symptoms | From baseline to 6 and 12 months of treatment
  Non Motor Symptoms Scale (NMSS) Total score and subdomains Cardiovascular, Sleep/Fatigue, Gastrointestinal, Urinary, Sexual functioning
Reason for transition to LCIG (or continuing oral therapy) | At Baseline, 6 and 12 month
  There are no data comparing long-term HRQL of LCIG versus peroral therapy
Change in participant's caregiver burden | From Baseline to 6 and 12 months of treatment
  Non Motor Symptoms Scale (NMSS) Total score and subdomains Cardiovascular, Sleep/Fatigue, Gastrointestinal, Urinary, Sexual functioning

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (27):
- Germany (23):
  - Universitaetsklinikum Aachen /ID# 204355, Aachen, North Rhine-Westphalia
  - Uniklinik Koln /ID# 148153, Cologne, North Rhine-Westphalia
  - Johannes Wesling Klin Minden /ID# 151481, Minden, North Rhine-Westphalia
  - KH Martha-Maria Halle Dolau /ID# 144634, Halle, Saxony-Anhalt
  - Klinikum Altenburger Land /ID# 139643, Altenburg
  - Kliniken Beelitz GmbH /ID# 144633, Beelitz-Heilstätten
  - Kupsch, Berlin, DE /ID# 144840, Berlin
  - Dr. Puzich, Berlin, DE /ID# 148226, Berlin
  - Delf, Berlin-Hoppegarten, DE /ID# 144632, Berlin-hoppengarten
  - Central Hospital Bremerhaven /ID# 144639, Bremerhaven
  - Neuro Centrum Odenwald /ID# 206998, Erbach im Odenwald
  - Herbst, Falkensee, DE /ID# 139642, Falkensee
  - Universitätsklinikum Freiburg /ID# 144640, Freiburg im Breisgau
  - Klinik Haag /ID# 137458, Haag
  - Wellach/Becker, Hamburg, DE /ID# 148228, Hamburg
  - Diak.hospital Henriettenstift /ID# 148222, Hanover
  - KH Agatharied /ID# 144636, Hausham
  - Klinikum Herford AdoeR /ID# 151482, Herford
  - Universitatsklinikum Jena_Duplicate /ID# 152813, Jena
  - Gertrudis-Klinik /ID# 144631, Leun-biskirchen
  - Universitatsklinikum Magdeburg /ID# 163197, Magdeburg
  - Philipps-Universitaet Marburg /ID# 116936, Marburg
  - Kliniken Berg /ID# 151484, Tübingen
- Switzerland (4):
  - University Hospital Zurich /ID# 153709, Zurich, Canton of Zurich
  - Luzerner Kantonsspital /ID# 153738, Lucerne
  - Klinik Bethesda /ID# 153739, Tschugg BE
  - Rehaklinik Zihlschlacht AG /ID# 153710, Zihlschlacht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/levodopa_carbidopa_P14-322.pdf